CLINICAL TRIAL: NCT02665455
Title: Evaluation of the Accuracy of the FreeStyle Libre Flash Glucose Monitoring System - Use in Pregnancy
Brief Title: FreeStyle Libre in Pregnancy Study
Acronym: FLIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADC-UK-VAL-15026
Record Dates: First submitted 2016-01-25; First posted 2016-01-27 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Sensing Technology
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): FreeStyle Libre Flash Glucose Monitoring System
  Interventions: Device: FreeStyle Libre Flash Glucose Monitoring System

INTERVENTIONS:
Device: FreeStyle Libre Flash Glucose Monitoring System — Subjects will wear the FreeStyle Libre Flash Glucose Monitoring System masked for 14 days.
  During these 14 days subjects will be asked to perform 4 blood glucose tests (pre-meals and before bedtime) per day. At the same time as the blood glucose test a sensor scan is performed.

SUMMARY:
To evaluate the point accuracy of the FreeStyle Libre Flash Glucose Monitoring System when used at home by pregnant women with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Type 1, type 2 or Gestational Diabetes Mellitus (GDM) (confirmed diagnosis via Oral Glucose Tolerance Test (OGTT))
* Currently testing Blood Glucose(BG), on average at least 2 times per day
* Participant is ≥12+0 weeks gestation with a singleton pregnancy
* In the investigator's opinion, technically capable of using device

Exclusion Criteria:

* Concomitant disease or condition that may compromise patient safety including and not limited to; cardiac disease or event, sickle cell disease, cystic fibrosis, severe mental illness, known or suspected eating disorder or any uncontrolled long term medical condition
* Currently receiving dialysis treatment or planning to receive dialysis during the study or, moderate to advanced nephropathy (serum creatinine ≥120 micromol/litre or total protein excretion exceeds 2 g/day or urinary albumin:creatinine ratio >30 mg/mmol, estimated glomerular filtration rate (eGFR) may not be used)
* Diabetic Ketoacidosis (DKA) (in the previous 6 months)
* Known (or suspected) allergy to medical grade adhesives
* In the investigator's opinion the participant is unsuitable to participate due to any other cause/reason, considering guidelines (e.g. National Institute for Health and Care Excellence (NICE) and International Diabetes Federation(IDF)) for Diabetes in Pregnancy for HbA1c and Blood Pressure
* Experiencing any of the following conditions for current pregnancy:

  * Pre-eclampsia
  * HELLP syndrome (haemolysis, elevated liver enzymes and low platelet count)
  * Prescribed Tocolytic drugs for treatment of preterm labour

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Austria (4):
  - VIVIT-Institut am Akad. Lehrkrankenhaus Feldkirch, Innere Medizin und Kardiologie, Feldkirch
  - Medizinische Universität Graz, Graz
  - Medizinische Universität Wien, Vienna
  - Krankenhaus Hietzing mit Neurologischem Zentrum Rosenhügel, Vienna
- United Kingdom (9):
  - Royal United Hospital, Bath
  - Southmead Hospital, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - St. James University Hospital, Leeds Teaching Hospitals NHS Trust, Leeds
  - Manchester Royal Infirmary, Manchester
  - James Cook University Hospital, Middlesbrough
  - John Radcliffe Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Warwick Hospital, Warwick

IPD SHARING:
Plan to Share IPD: No
Objective of study is to confirm accuracy of device in this patient population, so data cannot be shared with subjects until this is established

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eighty-three (83) participants were consented. Nine of the 83 participants withdrew from the study on or before Visit 1 and before the device was worn or used. All 74 participants that wore a sensor are included in the analysis.
Groups:
- Intervention: FreeStyle Libre Flash Glucose Monitoring System
  FreeStyle Libre Flash Glucose Monitoring System: Subjects will wear the FreeStyle Libre Flash Glucose Monitoring System masked for 14 days.
  During these 14 days subjects will be asked to perform 4 blood glucose tests (pre-meals and before bedtime) per day. At the same time as the blood glucose test a sensor scan is performed.
Period: Overall Study
Arm/Group | Intervention
Started | 83
Completed | 74
Not Completed | 9
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 83
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Point Accuracy Determined as % Within Consensus Error Grid Zone A
Description: Point accuracy of Sensor based glucose values versus fingerstick blood glucose determined as % within Consensus Error Grid zone A.
  Zone A is defined as the zone of "clinical accurate measurements with no effect on clinical action."
Time Frame: 14 days
Measure: Number (95% Confidence Interval); unit: percentage of results
Arm/Group | Intervention
Number analyzed (Participants) | 74
percentage of results | 88.1 [86 to 89.6]

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 3/83
Other Adverse Events (participants affected / at risk) | 0/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=83)
Pre eclampsia (Pregnancy, puerperium and perinatal conditions) | 2 (2) — None of the Serious Adverse Events are device related.
Vomiting & epigastric pain (Gastrointestinal disorders) | 1 (1) — None of the Serious Adverse Events are device related.
Decreased foetal movements (Pregnancy, puerperium and perinatal conditions) | 1 (1) — None of the Serious Adverse Events are device related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days